CLINICAL TRIAL: NCT03163134
Title: Lumbar Drain After Endoscopic Surgery of the Skull Base
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the fact data results were statistically significant among the two groups
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Paul Gardner, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO10030258
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-05

CONDITIONS: Quality of Life
Keywords: Lumbar Drain, CSF Leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- No Lumbar Drain Group (No Intervention): Group of patients that did not receive a lumbar drain after surgery
- Lumbar Drain Group (Experimental): Group of patients that received a lumbar drain after surgery
  Interventions: Device: Lumbar Drain

INTERVENTIONS:
Device: Lumbar Drain
  Arms: Lumbar Drain Group

SUMMARY:
The overall purpose of this study was to assess the necessity of lumbar drain placement after endoscopic endonasal approach (EEA) surgery in reducing cerebrospinal fluid (CSF) leak postoperatively and promote a standardization of its use.

DETAILED DESCRIPTION:
In the past, reconstructions were performed using fat grafts or fascia lata for EEA surgery. Considerably high postoperative CSF leaks were reported and were a major cause of concern due CSF fistula increasing risk of infection. Since external lumbar drain can lower CSF pressure and is believed to prevent post operative CSF leak, it was used commonly after EEA. With improvements in EEA skull base reconstructions using a nasal septal flap in the recent years, postoperative CSF leaks have been reported in much lower rates. With this improvement in reconstruction techniques, the use of lumbar drain may not be necessary as it may not significantly lower the risk of CSF leak further. In this prospective randomized study, we will randomize subjects at high risk for CSF leak to either receive a prophylactic lumbar drain or to not receive a prophylactic lumbar drain and compare the rate of CSF leaks and other complications in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients undergoing EEA for resection of brain tumors
* Dural defect greater than 1cm
* Extensive arachnoid dissection
* Dissection into a ventricle or cistern

Exclusion Criteria:

* Less than 18 years of age
* Spina Bifida

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2011-02-03 (Actual); Primary Completion 2015-04-27 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gardner, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zwagerman NT, Wang EW, Shin SS, Chang YF, Fernandez-Miranda JC, Snyderman CH, Gardner PA. Does lumbar drainage reduce postoperative cerebrospinal fluid leak after endoscopic endonasal skull base surgery? A prospective, randomized controlled trial. J Neurosurg. 2018 Oct 19;131(4):1172-1178. doi: 10.3171/2018.4.JNS172447. Print 2019 Oct 1. PMID 30485224

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult patients undergoing endoscopic endonasal approach (EEA) at the Center for Cranial Base Surgery of the University of Pittsburgh Medical Center from February 2011 to April 2015 were evaluated for enrollment.
Groups:
- Lumbar Drain Group: Group of patients that received a lumbar drain after surgery
  Lumbar Drain
Period: Overall Study
Arm/Group | No Lumbar Drain Group | Lumbar Drain Group
Started | 85 | 85
Completed | 85 | 85
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lumbar Drain Group: Group of patients that received a lumbar drain after surgery.
  Lumbar Drain
- Total: Total of all reporting groups
Arm/Group | No Lumbar Drain Group | Lumbar Drain Group | Total
Number analyzed (Participants) | 85 | 85 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (15.11) | 51 (15.49) | 52 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 56 | 105
  Male | 36 | 29 | 65
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 85 | 85 | 170

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cerebrospinal Fluid (CSF) Leak
Description: Determine the rate of CSF leak in endoscopic endonasal approach (EEA) patients who received lumbar drain placement and EEA patients who did not receive lumbar drain placement.
Time Frame: 1month
Measure: Count of Participants; unit: Participants
Arm/Group | No Lumbar Drain Group | Lumbar Drain Group
Number analyzed (Participants) | 85 | 85
Participants | 18 | 7
Statistical Analysis 1: Comparison: No Lumbar Drain Group vs Lumbar Drain Group; Test type: Other; p = 0.017, Chi-squared

2. Secondary Outcome: Number of Participants With Postoperative Complications
Description: Determine the rate of any postoperative complications related to Deep Vein Thrombosis (DVT), Pulmonary Embolism (PE), Meningitis and Respiratory infections in EEA patients who received lumbar drain placement and EEA patients who did not receive lumbar drain placement.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | No Lumbar Drain Group | Lumbar Drain Group
Number analyzed (Participants) | 85 | 85
Participants | 17 | 20
Statistical Analysis 1: Comparison: No Lumbar Drain Group vs Lumbar Drain Group; Test type: Other; p = 0.577, Chi-squared

ADVERSE EVENTS:
Time Frame: Three times a year
Arm/Group | No Lumbar Drain Group | Lumbar Drain Group
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes